CLINICAL TRIAL: NCT01229189
Title: Evaluation of the Effectiveness of Vitamin D Supplementation to Pregnant Women and Their Infants in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: John Snow, Inc. (Industry)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Professor and Founding Chair, Division of Women and Child Health, Aga Khan University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Vitamin D Study
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Vitamin D Deficiency; Pre Eclampsia; Stillbirths; Low Birth Weight; Prematurity
Keywords: Vitamin D; Effectiveness; Pregnant women and their neonates
MeSH Terms: conditions — Vitamin D Deficiency; Pre-Eclampsia; Stillbirth; Premature Birth | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maternal and Neonatal Intervention Arm (Experimental): Pregnant women will be individually randomized; a daily dose of vitamin D in 4000 IU will be given to Intervention group, started at 20-22 weeks of pregnancy till the time of delivery. The infants of this group will further stratify into two groups, one group will receive 400 IU of Vitamin D for 6 months as Intervention.
  Interventions: Dietary Supplement: Vitamin D
- Maternal and Neonatal Control Arm (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Maternal dose of 4000 IU daily for 20 weeks Neonatal dose of 400 IU daily for 24 weeks
  Arms: Maternal and Neonatal Intervention Arm
Dietary Supplement: Placebo — Placebo will be supplemented to pregnant women and their neonates in the same pattern as in intervention group.
  Arms: Maternal and Neonatal Control Arm

SUMMARY:
Vitamin D deficiency is wide spread in South Asian population and is contributing to burden of disease in this region including Pakistan. The relative importance of vitamin D deficiency, mutation in its receptor and maternal and child health has not been established in Pakistan and population based studies are required to explore and avert the maternal and Neonatal complications and consequences of Vitamin D deficiency

The trial will evaluate the effectiveness of Vitamin D supplementation to pregnant women and their Infants. It will be a double blind placebo controlled trial, which will be conducted in a rural district of Pakistan.

DETAILED DESCRIPTION:
The investigators are proposing a community based introduction of vitamin D supplementation and we intend to understand the complex relationship between vitamin D, the growth factors and maternal and infant anthropometric variables and hope to unravel the reasons of vitamin D deficiency in our population.

The investigators expect that if vitamin D is supplemented to pregnant women and their newborn infants it will inevitably replenish the micronutrient stores and aid to resolve the maternal and neonatal morbidity due to Vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women from 20-22 weeks of gestation and their infants, who will agree to take part in this study, will be enrolled.

Exclusion Criteria:

* Pregnant women with pre existing type 1 or type II diabetes
* Women with multiple fetuses, babies (twins, triplets)
* Pregnant women with high level of Vitamin D
* Babies with multiple congenital anomalies
* Babies with serious birth injury, birth asphyxia and serious infections
* Low birth weight less than 1.5
* Refuse to participate in the study

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 460 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Maternal and Neonatal complications | six months post enrolement
  Preeclampsia, hypertension ,poor weight gain etc during pregnancy.Still birth rates, Rate of low birth weight, prematurity,Neonatal seizures, Infants with growth failure, signs and symptoms of vitamin D deficiency. Infants with infections: pneumonia, diarrhea and Receptor polymorphism

SECONDARY OUTCOMES:
Prevalence and Risk factors for Maternal and Neonatal Vit D Deficiency | Six months post recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar A Bhutta, FRCPCH, PhD, Principal Investigator — Aga Khan University
Locations (1):
- Project Office Aga Khan University, Pind Dadan Khan, Punjab Province, Pakistan

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- See also: Official Website of the Aga Khan University — http://www.aku.edu